CLINICAL TRIAL: NCT02625454
Title: Randomized Control Trial of Intravenous Acetaminophen (OFIRMEV) for the Reduction of Intrapartum Maternal Fever and Fetal Tachycardia
Brief Title: Reduction of Intrapartum Fever With Intravenous Acetaminophen
Acronym: RIFIVA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Richmond University Medical Center (Other)
Responsible Party: Principal Investigator, Nisha Lakhi, MD, OBGYN Director of Research, Richmond University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015-09-06 RUMC
Record Dates: First submitted 2015-12-01; First posted 2015-12-09 (Estimated); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Fever; Oxidative Stress
Keywords: Acetaminophen; Labor; Intrapartum Fever; Maternal Fever; Fetal Tachycardia; Intravenous Acetaminophen
MeSH Terms: conditions — Fever | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intravenous Acetaminophen (Experimental): Subjects will receive 1000 mg of intravenous Acetaminophen q 6 hours, up to two doses and an oral placebo resembling oral acetaminophen
  Interventions: Drug: Intravenous Acetaminophen
- Oral Acetaminophen (Active Comparator): Subjects will receive 1000 mg of oral Acetaminophen q 6 hours, up to two doses and an intravenous placebo resembling intravenous acetaminophen
  Interventions: Drug: Oral Acetaminophen

INTERVENTIONS:
Drug: Intravenous Acetaminophen — 1000 mg Acetaminophen q 6 hours, given intravenously
  Other Names: OFIRMEV
  Arms: Intravenous Acetaminophen
Drug: Oral Acetaminophen — 1000 mg Acetaminophen q 6 hours given orally
  Other Names: Tylenol
  Arms: Oral Acetaminophen

SUMMARY:
The investigators plan to administer acetaminophen (Tylenol) for the treatment of fever in laboring patients by either an oral or intravenous (IV) route. The investigators want to see if the maternal fever will decrease faster with the IV or the oral dose. The investigators also want to look at other outcomes such as the cesarean section rate, the rate of neonatal intensive care unit admissions in both groups.

DETAILED DESCRIPTION:
This is a randomized, controlled, study of intravenous (IV) acetaminophen (OFIRMEV) versus orally administrated acetaminophen for the reduction of intrapartum maternal fever and fetal tachycardia. Compared to oral acetaminophen, intravenous acetaminophen has increased bioavailability and more rapid onset of action. IV acetaminophen has been used successfully in the management of fever in post-operative patients. Additionally, intravenous acetaminophen has also been used in the intrapartum setting for management of pain.However, the use of intravenous acetaminophen for the treatment of maternal temperature and subsequent fetal tachycardia, has not yet been evaluated.

The study will have two arms that will be randomized in a 1:1 ratio. A double dummy, double blind, comparator controlled study design will be utilized. After inclusion criteria have been satisfied, subjects in the control arm will receive an oral dose 1000 mg acetaminophen and an intravenous placebo resembling Ofirmev. The subjects in the experimental arm will receive 1000 mg of IV Ofirmev and an oral placebo resembling acetaminophen. Both groups will receive standard obstetrical care, continuous fetal monitoring, and antibiotics if there is suspected chorioamnionitis. The blinding technique will eliminate provider bias.

ELIGIBILITY:
Inclusion Criteria:

* Patients at Richmond University Medical Center that entered active labor (spontaneous or induced) and developed a systemic fever of greater than 38 degrees Celsius.

Exclusion Criteria:

* Exclusion Criteria: Infants delivered before 36 week gestation, stillbirths, congenital fetal anomalies, scheduled cesarean deliveries, and acetaminophen allergy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2016-12; Primary Completion 2019-05 (Actual); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Change in Maternal Body Temperature | 01, 15, 30, 60 and 90, 120, 180, 240, 300, 360 minutes following Time 01 (Time 01 = time when first dose of acetaminophen was administered

SECONDARY OUTCOMES:
Change in Fetal Heart Rate | 01, 15, 30, 60 and 90, 120, 180, 240, 300, 360 minutes following Time 01 (Time 01 = time when first dose of acetaminophen was administered
Mode of Delivery (cesarean section vs vaginal delivery) | Measured at point of delivery
Number of Cesarean Deliveries for Persistent Fetal Tachycardia | Measured at the point of delivery
Number of Patients with Diagnosis of Clinical Chorioamnionitis | Measured from admission to 7 days post-partum
Number of Patients with Diagnosis of Histological Chorioamnionitis | Measured from placenta histology collected at delivery
Neonatal Apgar Score | One and Five minutes of life
Number of Infants Admitted to Neonatal Intensive Care Unit | First 7 days of life
Number of Infants with Culture Positive Neonatal Sepsis | First 7 days of life
Number of infants requiring additional respiratory intervention | First 24 hours of life
Number of Infants Developing Neonatal Seizures | First 7 days of life
Number of infants with fetal acidosis | Point of Delivery
Maternal Levels of Pro-Inflammatory Mediators | Admission and 4 hours after delivery
  C-Reactive Protein (CRP), Tumor Necrosis Factor Alpha (TNF-α), Interleukin 6 (IL-6)
Levels of Pro-Inflammatory Mediator in Infant, collected from umbilical cord blood | Point of Delivery
  C-Reactive Protein (CRP), Tumor Necrosis Factor Alpha (TNF-α), Interleukin 6 (IL-6)
Maternal Levels of Oxidative Stress Markers | Admission and 4 hours after delivery
  Thioredoxin Reductase (TrxR), Gluathione (GSH)
Levels of Oxidative Stress Markers in Infant, collected from umbilical cord blood | point of delivery
  Thioredoxin Reductase (TrxR), Gluathione (GSH)
Levels of Acetaminophen in Cord Blood | point of delivery
Maternal Liver Function Test | 12-24 hours after delivery
  aspartate aminotransferase (AST), alanine aminotransferase (ALT)
Maternal White Blood Count (WBC) | Admission and 12-24 hours after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Nisha Lakhi, MD, Principal Investigator — Richmond University Medical Center
Locations (1):
- Richmond University Medical Center, Staten Island, New York, United States

REFERENCES:
- [Derived] Mehraban S, Nematian S, Mehraban SS, Petrucci S, Tricorico G, Parnas Z, Shats L, Kanninen T, Moretti M, Cabbad M, Lakhi N. Randomized control trial of intravenous acetaminophen for reduction of intrapartum maternal fever. Am J Obstet Gynecol MFM. 2021 Jan;3(1):100287. doi: 10.1016/j.ajogmf.2020.100287. Epub 2020 Dec 9. PMID 33451627